CLINICAL TRIAL: NCT01417325
Title: A Registry Study of Percutaneous Coronary Intervention Treatment in Beijing Area of P.R. China
Brief Title: Beijing Percutaneous Coronary Intervention Registry
Acronym: BJPCI Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yuejin Yang, Director of coronary heart disease center, vice president of Fuwai hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: Bciqcic-fw-01
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The registry study is to obtain the state of the art of the percutaneous coronary intervention state treatment for coronary heart disease in Beijing area of P.R.China in a real world. The data are collected from 48 hospitals in Beijing area using an uploading system through internet.

ELIGIBILITY:
Inclusion Criteria:

* Patients from selected 48 hospitals of Beijing, P.R.China
* Patients receiving coronal artery angiography or percutaneous coronary intervention therapy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients receiving coronal artery angiography or percutaneous coronary intervention therapy in selected 48 hospitals of Beijing, P.R.China.
Sampling Method: Non-Probability Sample
Enrollment: 700000 (Estimated)
Dates: Start 2010-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, doctor, Study Chair — Fuwai Heart Hospital & Cardiovascular Institute
Locations (1):
- Beijing cardiovascular intervention quality control and improvement center, Beijing, Beijing Municipality, China